CLINICAL TRIAL: NCT05277337
Title: A Phase IV, Randomized, Interventional, Study to Assess Subject Treatment Session Perception and Investigator Treatment Experience of Alluzience and Vacuum-Dried Botulinum Neurotoxin Type A for Aesthetic Use
Brief Title: Study Comparing Treatment With Alluzience vs Reconstituted Toxin
Acronym: STAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05PF2005; 2021-004748-62 (EudraCT Number)
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-06

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Alluzience) (Experimental): Single treatment at the baseline visit with Alluzience. Glabellar lines will be treated with 10 U/0.05 mL per injection point. In total 50 s.U in 0.25 mL for 5 injection points.
  Interventions: Biological: Alluzience
- Group 2 (powder BoNT-A: BOTOX/Vistabel) (Active Comparator): Single treatment at the baseline visit with powder BoNT-A (BOTOX/Vistabel). Glabellar lines will be treated with 4 U/0.1 mL per injection point. In total 20 U in 0.5 mL for 5 injection points.
  Interventions: Biological: powder BoNT-A (BOTOX/Vistabel)

INTERVENTIONS:
Biological: Alluzience — Botulinum Toxin Type A (BoNT-A) for treatment of glabellar lines; Mode of administration: intramuscular injection
  Arms: Group 1 (Alluzience)
Biological: powder BoNT-A (BOTOX/Vistabel) — Botulinum Toxin Type A (BoNT-A) for treatment of glabellar lines; Mode of administration: intramuscular injection
  Arms: Group 2 (powder BoNT-A: BOTOX/Vistabel)

SUMMARY:
This is a Phase IV, open-label, randomized, interventional, two-armed, multi-centre study to investigate subject treatment perception and Investigator treatment experience when using Alluzience or vacuum-dried botulinum neurotoxin type A (powder BoNT-A) for treatment of glabellar lines (GL).

DETAILED DESCRIPTION:
This is a Phase IV, open-label, randomized, interventional, two-armed, multi-centre study to investigate subject treatment perception and Investigator treatment experience when using Alluzience or vacuum-dried botulinum neurotoxin type A (powder BoNT-A) for treatment of glabellar lines (GL).

ELIGIBILITY:
Inclusion Criteria:

1. Female 18 to < 65 years of age.
2. Moderate to severe GL at maximum frown as assessed by the Investigator.
3. Female of non-childbearing potential (i.e., postmenopausal [absence of menstrual bleeding for 1 year prior to screening, without any other medical reason], or has undergone hysterectomy or bilateral oophorectomy). OR Female of childbearing potential with a negative urine pregnancy test at screening and baseline, and agrees to use a highly effective and approved contraceptive method for the duration of the study.
4. Time and ability to complete the study and comply with instructions.
5. Understands the study requirements and signed the informed consent form (ICF).
6. Subjects who have planned to undergo aesthetic facial treatment with powder toxin at the study site.
7. Previous use of any approved botulinum toxin in facial areas.

Exclusion Criteria:

1. Previous use of any botulinum toxin in facial area within 6 months prior to study treatment.
2. Female who is pregnant, breast feeding, or intends to conceive a child during the study.
3. Known allergy or hypersensitivity to any component of the study product or any botulinum toxin serotype.
4. Any known contraindication such as subject with bleeding disorder or subject currently using anticoagulants.
5. Previous use of any hyaluronic acid soft tissue augmentation therapy in the treated area within 3 months before baseline.
6. Previous soft tissue augmentation with any permanent (non-biodegradable such as silicone, polyacrylamide, etc) or semi-permanent (i.e., calcium hydroxylapatite, poly-L-Lactic acid or polymethyl-methacrylate) product; lifting threads, or autologous fat in the treatment area.
7. Subject has any prior or current psychiatric illness (e.g. Psychosis, depression, anxiety), alcohol or drug abuse, or is taking antidepressant, anxiolytic, or antipsychotic medication that, in the Investigator's opinion, could affect the subject's safety and/or participation in the study.
8. Other concurrent medical conditions, therapy, or other condition that, in the Investigator's opinion, would interfere with the evaluation of the study medication, safety or efficacy, and/or put the subject at risk if he/she participates in the study.
9. Participation in an investigational device or drug study within 30 days prior to study treatment or plans to enroll in any other investigational study during participation in this study.
10. Study site personnel, close relatives of the study site personnel (e.g. parents, children, siblings, or spouse), employees or close relatives of employees at the Sponsor company.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (3):
  - Galderma Research Site 2003, Bochum
  - Galderma Research Site 2001, Düsseldorf
  - Galderma Research Site 2002, Düsseldorf
- United Kingdom (5):
  - Galderma Research Site 1003, Edinburgh
  - Galderma Research Site 1004, London
  - Galderma Research Site 1006, London
  - Galderma Research Site 1001, London
  - Galderma Research Site 1002, Street

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chadha P, Gerber PA, Hilton S, Molina B, Haq S, Partridge J, Wong V, Hoffmann K, Persson C, Prygova I. Ready-to-use abobotulinumtoxinA solution versus powder botulinumtoxinA for treatment of glabellar lines: Investigators' and subjects' experience in a Phase IV study. J Cosmet Dermatol. 2024 Sep;23(9):2857-2866. doi: 10.1111/jocd.16359. Epub 2024 May 28. PMID 38807515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 centers in Germany and United kingdom from 04 February 2022 to 12 October 2022.
Pre-assignment Details: A total 153 participants were screened, of which 150 participants were randomized and enrolled, 99 participants in the Alluzience treatment group (Group 1) and 51 in the vacuum-dried botulinum neurotoxin type A (Powder BoNT-A) treatment group (Group 2).
Groups:
- Group 1 (Alluzience): Alluzience 0.25 mL single dose was administered as an intramuscular injection, through a syringe and needle at baseline visit (Day 0).
- Group 2 (Powder BoNT-A: BOTOX/Vistabel): Powder BoNT-A 0.5 mL single dose was administered as an intramuscular injection, through a syringe and needle at baseline visit (Day 0).
Period: Overall Study
Arm/Group | Group 1 (Alluzience) | Group 2 (Powder BoNT-A: BOTOX/Vistabel)
Started | 99 | 51
Completed | 96 | 51
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 2 (Powder BoNT-A: BOTOX/Vistabel): Injection Powder BoNT-A 0.5 mL single dose was administered as an intramuscular injection, through a syringe and needle at baseline visit (Day 0).
- Total: Total of all reporting groups
Arm/Group | Group 1 (Alluzience) | Group 2 (Powder BoNT-A: BOTOX/Vistabel) | Total
Number analyzed (Participants) | 99 | 51 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (10.27) | 44.6 (10.91) | 45.4 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 51 | 150
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 96 | 46 | 142
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 94 | 49 | 143
  Race: Black or African American | 1 | 1 | 2
  Race: Asian | 1 | 1 | 2
  Race: Other Asian | 2 | 0 | 2
  Race: Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time Needed to Prepare Alluzience and Powder BoNT A
Description: Time to prepare Alluzience and powder Bont A according to protocol was reported.
Time Frame: Baseline (Day 0)
Population: The full analysis set (FAS) population included all randomized and treated participants.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (Alluzience) | Group 2 (Powder BoNT-A: BOTOX/Vistabel)
Number analyzed (Participants) | 99 | 51
Minutes | 0.55 (0.414) | 1.57 (0.831)

2. Secondary Outcome: Percentage of Participants Injected With Alluzience for Whom Investigator Did Not Face Technical Issue/Problems When Using a Ready-to-use Product as Compared to a Product to be Reconstituted
Description: Percentage of participants injected with Alluzience for whom investigator did not face technical issue/problems when using a ready-to-use product as compared to a product to be reconstituted, assessed using answers within each answer option (strongly agree, agree, neither agree nor disagree, disagree and strongly disagree) was reported.
Time Frame: Baseline (Day 0)
Population: The full analysis set (FAS) population included all randomized and treated participants.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 (Alluzience)
Number analyzed (Participants) | 99
percentage of participants
  Strongly Agree | 91.9
  Agree | 8.1

3. Secondary Outcome: Percentage of Participants Injected With Powder Bont-A for Whom Investigator Experienced Issues While Reconstitution
Description: Percentage of participants injected with Powder Bont-A for whom investigator experienced issues while reconstitution was assessed using a questionnaire (Yes/No). Percentage of participants with answer "Yes" was reported.
Time Frame: Baseline (Day 0)
Population: The full analysis set (FAS) population included all randomized and treated participants.
Measure: Number; unit: percentage of participants
Arm/Group | Group 2 (Powder BoNT-A: BOTOX/Vistabel)
Number analyzed (Participants) | 51
percentage of participants | 2

4. Secondary Outcome: Investigator Treatment Session Questionnaire
Description: Treating investigators who injected participant with Alluzience answered questions 1 through 12 of the investigator treatment questionnaire for each participant at baseline. The options for each question were strongly agree, agree, neither agree nor disagree, disagree and strongly disagree.
Time Frame: Baseline (Day 0)
Population: The full analysis set (FAS) population included all randomized and treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Alluzience)
Number analyzed (Participants) | 99
Participants
  Prefer to utilize ready-to-use product than reconstituted product: Strongly Agree/Agree | 80
  Prefer to utilize ready-to-use product than reconstituted product: Neither Agree nor Disagree | 19
  Prefer to utilize ready-to-use product than reconstituted product: Disagree/Strongly disagree | 0
  Gave more time to explain treatment procedure using ready-to-use product than reconstituted product: Strongly Agree/Agree | 96
  Gave more time to explain treatment procedure using ready-to-use product than reconstituted product: Neither Agree nor Disagree | 2
  Gave more time to explain treatment procedure using ready-to-use product than reconstituted product: Disagree/Strongly disagree | 1
  Could save time on the reconstitution and injection procedure to do something else: Strongly Agree/Agree | 92
  Could save time on the reconstitution and injection procedure to do something else: Neither Agree nor Disagree | 7
  Could save time on the reconstitution and injection procedure to do something else: Disagree/Strongly disagree | 0
  Felt more relaxed/less stressed in not having to reconstitute the product to be injected: Strongly Agree/Agree | 68
  Felt more relaxed/less stressed in not having to reconstitute the product to be injected: Neither Agree nor Disagree | 24
  Felt more relaxed/less stressed in not having to reconstitute the product to be injected: Disagree/Strongly disagree | 7
  Feel more secure with pre-diluted solution and don't have to reconstitute the product myself: Strongly Agree/Agree | 64
  Feel more secure with pre-diluted solution and don't have to reconstitute the product myself: Neither Agree nor Disagree | 25
  Feel more secure with pre-diluted solution and don't have to reconstitute the product myself: Disagree/Strongly disagree | 10
  Have a good feeling about injecting a modern and innovative product than reconstituted product: Strongly Agree/Agree | 81
  Have a good feeling about injecting a modern and innovative product than reconstituted product: Neither Agree nor Disagree | 17
  Have a good feeling about injecting a modern and innovative product than reconstituted product: Disagree/Strongly disagree | 1
  More precise in my injection with a ready-to-use product than reconstituted product: Strongly Agree/Agree | 75
  More precise in my injection with a ready-to-use product than reconstituted product: Neither Agree nor Disagree | 12
  More precise in my injection with a ready-to-use product than reconstituted product: Disagree/Strongly disagree | 12
  Like to propose new innovative treatment with liquid ready-to-use product to my patient: Strongly Agree/Agree | 86
  Like to propose new innovative treatment with liquid ready-to-use product to my patient: Neither Agree nor Disagree | 11
  Like to propose new innovative treatment with liquid ready-to-use product to my patient: Disagree/Strongly disagree | 2
  Produced less waste of non-toxin material using ready-to-use product than reconstituted product: Strongly Agree/Agree | 96
  Produced less waste of non-toxin material using ready-to-use product than reconstituted product: Neither Agree nor Disagree | 3
  Produced less waste of non-toxin material using ready-to-use product than reconstituted product: Disagree/Strongly disagree | 0
  When I use a ready-to-use toxin I spend less materials for injection: Strongly Agree/Agree | 98
  When I use a ready-to-use toxin I spend less materials for injection: Neither Agree nor Disagree | 1
  When I use a ready-to-use toxin I spend less materials for injection: Disagree/Strongly disagree | 0
  Believe that the use of ready-to-use toxin is better for the environment as I produce less waste: Strongly Agree/Agree | 99
  Believe that the use of ready-to-use toxin is better for the environment as I produce less waste: Neither Agree nor Disagree | 0
  Believe that the use of ready-to-use toxin is better for the environment as I produce less waste: Disagree/Strongly disagree | 0
  Feel more confident when injecting a product free from animal and human excipients: Strongly Agree/Agree | 82
  Feel more confident when injecting a product free from animal and human excipients: Neither Agree nor Disagree | 17
  Feel more confident when injecting a product free from animal and human excipients: Disagree/Strongly disagree | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from treatment until the end of the participant's participation ( for Alluzience upto 6 months and BOTOX upto 1 month)
Description: The safety population was to include all participants who were administered study product.
Arm/Group | Group 1 (Alluzience) | Group 2 (Powder BoNT-A: BOTOX/Vistabel)
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/51
Other Adverse Events (participants affected / at risk) | 18/99 | 0/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Alluzience) (N=99) | Group 2 (Powder BoNT-A: BOTOX/Vistabel) (N=51)
Injecttion Site Pain (General disorders) | 11 | 0
Injection Site Haematoma (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Tension headache (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agree not to present/publish any data or reports collected individually or by subgroup of trial sites prior to first publication based on data obtained from all sites. Investigators can publish results 18 months after the completion of the trial, but Sponsor shall have the right to review any proposed publication before publication/presentation to prevent the disclosure of confidential information. Sponsor can refuse the publication, delay it or request amendment of its contents

DOCUMENTS (2):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT05277337/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT05277337/SAP_001.pdf